CLINICAL TRIAL: NCT01759407
Title: A Prospective, Double-blinded, Randomized Comparison of Ultrasound-guided Femoral Nerve Block With Lateral Femoral Cutaneous Nerve Block Versus Standard Anesthetic Management for Traumatic Femur Fracture Repair in the Pediatric Population
Brief Title: Femoral Nerve Block for Femur Fracture Repair in Pediatrics
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis showed no significant difference between study arms.
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Nicole Elsey, Clinical Assistant Professor, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB16-00338
Record Dates: First submitted 2012-12-29; First posted 2013-01-03 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Traumatic Femur Fracture
MeSH Terms: interventions — Ropivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral Nerve Block (Active Comparator): Ropivicaine 0.2% with epinephrine 1:200,000 will be used for patients between 10kg and up to 25kg in weight; ropivicaine 0.5% with epinephrine 1:200,000 will be used for patients greater than or equal to 25kg
  Interventions: Drug: Ropivicaine; Drug: Epinephrine
- Standard Anesthetic Management (No Intervention)

INTERVENTIONS:
Drug: Ropivicaine
  Other Names: Naropin
  Arms: Femoral Nerve Block
Drug: Epinephrine
  Arms: Femoral Nerve Block

SUMMARY:
The purpose of this study is to prospectively compare post-operative pain relief in pediatric patients undergoing traumatic femur fracture repair who have received either a femoral nerve block with a lateral femoral cutaneous nerve block or a standard anesthetic for analgesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II
* Weight greater than or equal to 10kg
* Presenting for repair of traumatic femur fracture

Exclusion Criteria:

* ASA physical status > II
* Co-morbid diseases (cardiac, pulmonary, neurological disease)
* Patients having concomitant procedures
* Abnormal neurovascular examination in the injured leg
* Presence of vascular compromise in the affected lower extremity
* Mechanism of sustained injury via crush injury
* Use of therapeutic dose anticoagulants or presence of a bleeding disorder

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2013-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Elsey, MD, Principal Investigator — Nationwide Children's
Locations (1):
- Nationwide Children's, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Femoral Nerve Block: Ropivicaine 0.2% with epinephrine 1:200,000 will be used for patients between 10kg and up to 25kg in weight; ropivicaine 0.5% with epinephrine 1:200,000 will be used for patients greater than or equal to 25kg
  Ropivicaine
Period: Overall Study
Arm/Group | Femoral Nerve Block | Standard Anesthetic Management
Started | 10 | 9
Completed | 10 | 7
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Femoral Nerve Block | Standard Anesthetic Management | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.1 (3.5) | 7.7 (3.4) | 8 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Post-anesthesia Care Unit (PACU) Pain Scores
Description: Hannallah et al developed the Objective Pain Scale (OPS) to monitor pain in children after surgery. Parameters: (1) systolic blood pressure, (2) crying, (3) movement, (4) agitation (confused, excited), (5) complains of pain (may not be possible in younger children). Interpretation: minimum score: 0; maximum score: 10; maximum score if too young to complain of pain: 8; the higher the score, the greater the degree of pain.
Time Frame: 30 mins after surgery
Measure: Median (Inter-Quartile Range); unit: pain score
Arm/Group | Femoral Nerve Block | Standard Anesthetic Management
Number analyzed (Participants) | 10 | 7
pain score | 0 [0 to 0] | 3 [0 to 4]

2. Secondary Outcome: Intraoperative End-tidal Isoflurane %
Description: Median end-tidal isoflurane concentration per participant during the average 1 1/2 hr. surgery.
Time Frame: 1 1/2 hr.
Measure: Median (Inter-Quartile Range); unit: percentage of isoflurane
Arm/Group | Femoral Nerve Block | Standard Anesthetic Management
Number analyzed (Participants) | 10 | 7
percentage of isoflurane | 1.1 [1.0 to 1.4] | 1.5 [1.0 to 1.7]

3. Secondary Outcome: Time to First Opioid Dose
Description: Median time between PACU discharge and first opioid dose on the ward.
Time Frame: From PACU discharge until first opioid dose on the ward, assessed up to 24 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Femoral Nerve Block | Standard Anesthetic Management
Number analyzed (Participants) | 10 | 7
hours | 3.3 [2.8 to 5.3] | 3.8 [2.9 to 8.1]

ADVERSE EVENTS:
Arm/Group | Femoral Nerve Block | Standard Anesthetic Management
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes